CLINICAL TRIAL: NCT00961805
Title: Effectiveness of Dance on Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Andreia Salvador Baptista, Federal Unversity of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1044/06
Record Dates: First submitted 2009-04-30; First posted 2009-08-19 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Treatment; Dance; Randomized controlled study; Exercise
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dance Group (Experimental): Belly dance
  Interventions: Behavioral: Dance
- Control Group (No Intervention): Waiting list
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Dance — Belly dance classes twice a week for 16 weeks. Each class had a maximum of eight students. The classes were administered by a physiotherapist with eight years of experience in belly dance. Classes began with a warm-up exercise, followed by the predetermined movements for the day, choreography and a cool-down exercise. The participants received a compact disc with music and an exercise book with the history and movements proposed for the program. Beginning in the fourth week, a set sequence of movements in the form of choreography was established for memorization and training at home.
  Arms: Dance Group
Other: Control Group — The control group did not receive any intervention. They attended all assessments and remained on the waiting lis (after the end of the study was offered to this group the same treatment in the intervention group).
  Arms: Control Group

SUMMARY:
The aim of the present study is to assess the effectiveness of belly dance as a treatment for pain and improving the quality of life of patients with fibromyalgia.

Eighty female patients with fibromyalgia between 18 to 65 years were randomly allocated to a dance group (n=40) and control group (n=40). Patients in the dance group underwent 16 weeks of belly dance twice a week, while the patients in the control group remained on a waiting list. Patients were evaluated with regard to pain (Visual Analogue Scale), function (6 minute walk test), quality of life (Fibromyalgia Impact Questionnaire and SF-36), depression (Beck Inventory), anxiety (State-Trait Anxiety Inventory) and self-image (Body Dysmorphic Disorder Examination) questionnaire. Evaluations were carried out at baseline, after 16 weeks and after 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* classification of fibromyalgia based on the criteria of the American College of Rheumatology
* female gender
* aged between 18 and 65 years

Exclusion Criteria:

* not having altered treatment in previous three years
* having signed a term of informed consent
* patients with other rheumatic diseases, painful osteoarticular conditions, uncontrolled cardiopulmonary disease, diseases of the lower limbs or uncontrolled diabetes were excluded

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreia S Baptista, PT, Principal Investigator — Federal University of São Paulo; Jamil Natour, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Baptista AS, Villela AL, Jones A, Natour J. Effectiveness of dance in patients with fibromyalgia: a randomized, single-blind, controlled study. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):18-23. Epub 2012 Dec 14. PMID 23020850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of patients started in August 2007 and finished in April 2008. The recruitment was made in Sao Paulo Hospital division of Rheumatology
Groups:
- Dance Group: The participants in the dance group took one-hour belly dance classes twice a week for 16 weeks. Each class had a maximum of eight students. The classes were administered by a physiotherapist with eight years of experience in belly dance. Classes began with a warm-up exercise, followed by the predetermined movements for the day, choreography and a cool-down exercise. The participants received a compact disc with music and an exercise book with the history and movements proposed for the program. Beginning in the fourth week, a set sequence of movements in the form of choreography was established for memorization and training at home.
Period: Overall Study
Arm/Group | Control Group | Dance Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group Control: The waiting list
- Total: Total of all reporting groups
Arm/Group | Group Control | Dance Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.5) | 49.5 (10.9) | 49.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale for Pain
Description: score between 0 and 100 where 0 is no pain and 100 in unbearable pain
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
mm
  Baseline | 75 (13) | 75 (17)
  After 16 weeks | 75 (14) | 46 (20)
  After 32 weeks | 73 (17) | 47 (26)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Sample size was calculated by visual analogue scale for pain (alpha error of 5%, beta error of 20% and standard deviation of 2). The sample was determined to contain 30 patients in each group. Ten additional patients were added to compensate possible losses. Analysis was intention to treat using the LOCF technique; Test type: Superiority or Other; p < 0.001, ANOVA — Differences in the behavior of the groups over time

2. Secondary Outcome: Function - 6 Minute Walk Test
Description: meters traveled on a 20-meter course over a six-minute period
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
meters
  Baseline | 332 (66.7) | 372.8 (80.2)
  after 16 weeks | 344.3 (72.7) | 443.5 (78.3)
  after 32 weeks | 343 (77.9) | 431 (88.7)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p < 0.001, ANOVA — Differences in the behavior of the groups over time

3. Secondary Outcome: Quality of Life - Fibromyalgia Impact Questionnaire
Description: score between 0 from 10 with 0 indicating no impairment and 10 indicating maximum impairment
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 6.34 (1.29) | 5.89 (1.39)
  After 16 weeks | 6.61 (1.53) | 4.69 (1.73)
  After 32 weeks | 5.9 (1.86) | 4.26 (1.81)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p < 0.003, ANOVA — Differences in the behavior of the groups over time

4. Secondary Outcome: Quality of Life - SF-36 -Functional Capacity
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 32.6 (18.9) | 44.9 (18.9)
  After 16 weeks | 33.1 (18.6) | 52.9 (21.1)
  After 32 weeks | 39.1 (22) | 56.3 (19.9)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.146, ANOVA — Differences in the behavior of the groups over time

5. Secondary Outcome: Quality of Life - SF-36 - Physical Limitation
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 8.8 (17.9) | 24.7 (32.2)
  After 16 weeks | 10.4 (21.6) | 40.5 (30.6)
  After 32 weeks | 13.8 (26.5) | 36.5 (13.8)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.131, ANOVA — Differences in the behavior of the groups over time

6. Secondary Outcome: Quality of Life - Sf-36 - Pain
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 25.7 (13.4) | 29.6 (17.5)
  After 16 weeks | 25.1 (14.2) | 44.7 (20.7)
  After 32 weeks | 29.1 (21.1) | 46 (19.2)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p < 0.001, ANOVA — Differences in the behavior of the groups over time

7. Secondary Outcome: Quality of Life - Sf-36 - General Health State
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 38 (16.5) | 46 (21.7)
  After 16 weeks | 38.1 (18.3) | 45 (21.3)
  After 32 weeks | 41.5 (21.4) | 44.9 (15.6)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.580, ANOVA — Differences in the behavior of the groups over time

8. Secondary Outcome: Quality of Life - SF-36 - Vitality
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 29 (18.2) | 41.3 (18.8)
  After 16 weeks | 30.7 (18.1) | 50 (22.8)
  After 32 weeks | 37.1 (21.8) | 47.6 (24.5)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.082, ANOVA — Differences in the behavior of the groups over time

9. Secondary Outcome: Quality of Life - SF-36 - Social Aspects
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 47.6 (23.1) | 52.6 (27.7)
  After 16 weeks | 47.6 (24.5) | 64.1 (28)
  After 32 weeks | 51.3 (25.5) | 57.2 (27)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.055, ANOVA — Differences in the behavior of the groups over time

10. Secondary Outcome: Quality of Life - SF-36 - Emotional Aspects
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 21.2 (33.1) | 34.2 (36.9)
  After 16 weeks | 17.5 (26.1) | 55 (33.6)
  After 32 weeks | 31.5 (38.7) | 51.9 (39.6)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.003, ANOVA — Differences in the behavior of the groups over time

11. Secondary Outcome: Quality of Life - SF-36 - Mental Health
Description: score between 0 from 100, with higher scores denoting better quality of life
Time Frame: baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 43.4 (24) | 46 (19.9)
  After 16 weeks | 44.5 (26.6) | 54.2 (20.7)
  After 32 weeks | 46.2 (22.6) | 52.3 (20.8)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.021, ANOVA — Differences in the behavior of the groups over time

12. Secondary Outcome: Depression - Beck Inventory
Description: score between 0 from 63, with higher score indicating greater depression
Time Frame: Baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 21.2 (13) | 23.9 (14.7)
  After 16 weeks | 23.5 (11.5) | 20.2 (13.2)
  After 32 weeks | 23.5 (13.7) | 23.1 (15.3)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.136, ANOVA — Differences in the behavior of the groups over time

13. Secondary Outcome: Self-image - Body Dysmorphic Disorder Examination Questionnaire
Description: scored between 0 from 168, with higher scores indicating greater level of dissatisfaction with self-image
Time Frame: Baseline, after 16 weeks and after 32 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Dance Group
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 48.8 (34.2) | 42.8 (32.6)
  After 16 weeks | 50.5 (29.4) | 33.6 (25.9)
  After 32 weeks | 46.9 (31.8) | 41.1 (24.4)
Statistical Analysis 1: Comparison: Control Group vs Dance Group; Test type: Superiority or Other; p = 0.009, ANOVA — Differences in the behavior of the groups over time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No